CLINICAL TRIAL: NCT02825797
Title: An Phase 1b Study of the Safety, Pharmacokinetics and Antiretroviral Activity of the Combination of 3BNC117 and 10-1074 in HIV-infected Individuals
Brief Title: 3BNC117 and 10-1074 in HIV-infected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCA-0906
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Broadly neutralizing antibody; 3BNC117; 10-1074
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — 3BNC117 antibody; Antibodies, Monoclonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (5):
- Group 1A (Experimental): HIV-infected individuals, on ART with HIV-1 RNA < 20 copies/ml will be randomized in a 2:1 ratio to receive one intravenous infusion of 3BNC117 and one intravenous infusion of 10-1074), each dosed at 10 mg/kg OR placebo (sterile saline), on day 0.
  Interventions: Drug: 3BNC117; Drug: 10-1074; Drug: Placebo
- Group 1B (Experimental): HIV-infected individuals, on ART with HIV-1 RNA < 20 copies/ml will be randomized in a 2:1 ratio to receive one intravenous infusion of 3BNC117 and one intravenous infusion 10-1074, each dosed at 30 mg/kg, OR placebo (sterile saline), on day 0.
  Interventions: Drug: 3BNC117; Drug: 10-1074; Drug: Placebo
- Group 1C (Experimental): HIV-infected individuals, off ART will be administered one infusion of 3BNC117 and one infusion 10-1074, each dosed at 30 mg/kg, on day 0.
  Interventions: Drug: 3BNC117; Drug: 10-1074
- Group 2 (Experimental): HIV-infected individuals, on ART with HIV-1 RNA < 20 copies/ml will be administered three infusions of 3BNC117 and three infusions of 10-1074, each dosed at 30 mg/kg, on days 0, 21 and 42. Participants enrolled in Group 2 will undergo an analytical treatment interruption and they will discontinue their antiretroviral (ART) regimen on day 2.
  Interventions: Drug: 3BNC117; Drug: 10-1074; Other: Analytical treatment interruption
- Group 3 (Experimental): HIV-infected individuals, off ART who will be administered three infusions of 3BNC117 and three infusions of 10-1074, each dosed at 30 mg/kg on days 0, 14 and 28.
  Interventions: Drug: 3BNC117; Drug: 10-1074

INTERVENTIONS:
Drug: 3BNC117 — Intravenous infusion of 3BNC117
  Other Names: Monoclonal Antibody
Drug: 10-1074 — Intravenous infusion of 10-1074
  Other Names: Monoclonal Antibody
Other: Analytical treatment interruption — Analytical treatment interruption
  Other Names: ART interruption
  Arms: Group 2
Drug: Placebo — Intravenous infusion of placebo (sterile saline)
  Other Names: Sterile Saline
  Arms: Group 1A; Group 1B

SUMMARY:
This is a phase 1b clinical trial to evaluate the safety, pharmacokinetics and the antiretroviral effects of the combination of two anti-human immunodeficiency virus (HIV) broadly neutralizing antibodies, 3BNC117 and 10-1074, administered intravenously in HIV-infected individuals. This study is intended to support the development of the combination of 3BNC117 and 10-1074 mAbs for use in the treatment of HIV-1 infection.

DETAILED DESCRIPTION:
The proposed study is a Phase 1b clinical trial to evaluate the safety, pharmacokinetics and the antiretroviral effects of the combination of two anti-HIV broadly neutralizing antibodies, 3BNC117 and 10-1074, administered intravenously in HIV-infected individuals.

The study includes 5 study groups. Study participants will be administered one or three intravenous infusions of 3BNC117 and 10-1074, each mAb dosed at 10 or 30 mg/kg:

Single dose groups:

Group 1A (n=6) - HIV-infected individuals, on antiretroviral therapy (ART) with HIV-1 RNA < 20 copies/ml will be randomized in a 2:1 ratio to receive one intravenous infusion of 3BNC117 and one infusion of 10-1074, each dosed at 10 mg/kg (n=4), OR placebo (sterile saline; n=2), on day 0.

Group 1B (n=6) - HIV-infected individuals, on ART with HIV-1 RNA < 20 copies/ml will be randomized in a 2:1 ratio to receive one intravenous infusion of 3BNC117 and one infusion 10-1074, each dosed at 30 mg/kg (n=4), OR placebo (sterile saline; n=2), on day 0.

Participants and investigators will be blinded to study assignment in groups 1A and 1B.

Group 1C (n=4) - HIV-infected individuals, off ART will be administered one infusion of 3BNC117 and one infusion 10-1074, each dosed at 30 mg/kg, on day 0.

Three doses groups:

Group 2 (n=15) - HIV-infected individuals, on ART who will be administered three infusions of 3BNC117 and three infusions of 10-1074, each dosed at 30 mg/kg, on days 0, 21 (week 3) and 42 (week 6). Participants enrolled in Group 2 will discontinue their antiretroviral (ART) regimen on day 2.

Group 3 (n=6) - HIV-infected individuals, off ART who will be administered three infusions of 3BNC117 and three infusions of 10-1074, each dosed at 30 mg/kg on days 0, 14 (week 2) and 28 (week 4).

Following 3BNC117 and 10-1074 infusions, study participants will return for safety assessments at multiple time points. Blood samples will be collected for safety testing at weeks 1, 2, and 4 following each mAb infusion, then bi-monthly or monthly until the end of study follow up.

Serum samples for PK (pharmacokinetic) measurements will be collected before the start of the first mAb infusion. Peak PK sampling for 3BNC117 will occur following the completion of the 3BNC117 infusion and prior to the start of the 10-1074 infusion. Peak PK sampling for 10-1074 will occur following the completion of the 10-1074 infusion. Additional samples for PK assessments will be collected at multiple time points during study follow up.

Samples will also be collected for measurement of HIV-1 plasma RNA levels before 3BNC117 and 10-1074 infusions (screen, pre-infusion and day 0), at all follow up visits in Groups 1A, 1B and 2, and weekly during the ATI period and at later time points in Group 2.

All participants will be followed for 24 weeks after the last 3BNC117 and 10-1074 infusions.

ELIGIBILITY:
Inclusion Criteria:

All groups:

* Age 18 to 65.
* HIV-1 infection confirmed by two independent laboratory assays.
* If sexually active male or female, and participating in sexual activity that could lead to pregnancy, agrees to use two effective methods of contraception (i.e. condom with spermicide, diaphragm with spermicide, hormone-eluting intrauterine device (IUD), hormone-based contraceptive with condom) for the study duration.

Groups 1A and 1B:

* HIV-infected volunteers on ART with HIV-1 plasma RNA levels < 20 copies/ml.
* Current CD4 cell count > 300 cells/μl.

Groups 1C and 3:

* HIV-infected volunteers off ART with detectable HIV-1 plasma RNA levels < 100,000 copies/ml by standard assays.
* Current CD4 cell count > 300 cells/μl.

Group 2:

* On antiretroviral therapy for a minimum of 24 months, with plasma HIV-1 RNA levels of < 50 copies/ml for at least 18 months, and < 20 copies/ml at screening. Note: a single viral load measurement > 50 but < 500 copies/ml during this time period is allowed.
* Current CD4+ T cell counts > 500 cells/μl. CD4 cell count nadir > 200 cells/μl.
* If on an NNRTI-based regimen willing to switch to a dolutegravir-based regimen for 4 weeks prior to discontinuing ART.

Exclusion Criteria:

* Have a history of AIDS-defining illness within 3 year prior to enrollment.
* History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
* Any clinically significant acute or chronic medical condition (such as autoimmune diseases or coronary artery disease), other than HIV infection, that in the opinion of the investigator would preclude participation.
* Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood.
* History of resistance to 2 or more classes of antiretroviral medication or known resistance to dolutegravir in participants on non-nucleoside reverse-transcriptase inhibitors (NNRTI), who would switch regimen prior to ATI (Group 2).
* Laboratory abnormalities in the parameters listed below:
* Absolute neutrophil count ≤ 1,000 cells/l
* Hemoglobin ≤ 10 gm/dL
* Platelet count ≤ 100,000 cells/l
* Alanine Aminotransferase (AST) ≥ 1.5 x ULN
* Aspartate Aminotransferase (AST) ≥ 1.5 x ULN
* Alkaline phosphatase ≥ 1.5 x ULN
* Total bilirubin > 1.0 ULN
* eGFR < 60 mL/min/1.73m2
* Pregnancy or lactation;
* Any vaccination within 14 days prior to 3BNC117 and 10-1074 administration;
* Subjects with known hypersensitivity to any constituent of the investigational products;
* Receipt of any therapeutic HIV vaccine or monoclonal antibody therapy of any kind in the past;
* Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
The number of participants with adverse events 1 week after 3BNC117 and 10-1074 infusions in all study groups. | 1 week following each combination of 3BNC117 and 10-1074 infusion
  Adverse events include: signs, symptoms and laboratory abnormalities, in addition to local and systemic reactogenicity
The decline in plasma HIV-1 RNA levels by a standard clinical assay in participants off ART enrolled in groups 1C and 3. | 20-24 weeks
The percentage of participants who meet ART re-initiation criteria (plasma HIV-1 RNA ≥ 200 copies/ml and/or CD4 count < 350 cells/μl on two consecutive measurements) prior to 8 weeks after ART interruption in group 2. | 30 weeks
Time to meeting ART re-initiation criteria (plasma HIV-1 RNA level ≥ 200 copies/ml, CD4+ T cell count < 350 cells/l in 2 consecutive measurements) following ART interruption in group 2. | 30 weeks

SECONDARY OUTCOMES:
The number of participants with adverse events that occur during study follow up after 3BNC117 and 10-1074 infusions in all study groups. | 20-30 weeks
  Adverse events include signs, symptoms and laboratory abnormalities.
The serum level of 3BNC117 and 10-1074 at the time of viral rebound in all study groups. | 20-30 weeks
Number of participants with induced anti-3BNC117 and anti-10-1074 antibodies. | 20-30 weeks
Level of induced anti-3BNC117 and anti-10-1074 antibodies. | 20-30 weeks
Change in number of CD4+ T cells/uL | 20-30 weeks

OTHER OUTCOMES:
Changes in viral envelope sequences following 3BNC117 and 10-1074 infusions (groups 1C, 2-3) | 20-30 weeks
Phylogenetic comparison of viruses grown from PBMCs collected from subjects while on ART to rebound viruses collected after treatment interruption (group 2). | 20-30 weeks
Levels of cell-associated HIV-1 RNA and DNA before and after 3BNC117 and 10-1074 infusions in HIV-infected individuals. | 20-30 weeks
Analysis of HIV-1 integration sites before and after 3BNC117 and 10-1074 infusions in HIV-infected individuals. | 20-30 weeks
HIV-1 specific T and B immune responses following 3BNC117 and 10-1074 infusions (groups 1-3). | 20-30 weeks
  These will be measured by intracellular cytokine staining and by TZM.bl assays against a panel of viruses from multiple HIV clades.
Elimination half-life (t1/2) of 3BNC117 and 10-1074 | 20-30 weeks
Clearance (CL/F) of 3BNC117 and 10-1074 | 20-30 weeks
Volume of distribution (Vz/F) of 3BNC117 and 10-1074 | 20-30 weeks
Area under the plasma concentration versus time curve (AUC) of 3BNC117 and 10-1074 | 20-30 weeks
Decay Curves of 3BNC117 and 10-1074 | 20-30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — Rockefeller University
Locations (2):
- The Rockefeller University, New York, New York, United States
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No